CLINICAL TRIAL: NCT07034261
Title: Continuous Glucose Monitoring to Detect Postpartum Dysglycemia in Patients With Gestational Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB25-0910
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Gestational Diabetes
Keywords: CGM Device
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Blinded Continuous Glucose Monitoring Device (Experimental): Subjects will wear a blinded continuous glucose monitoring device.
  Interventions: Device: Blinded Continuous Glucose Monitoring Device

INTERVENTIONS:
Device: Blinded Continuous Glucose Monitoring Device — Subjects will be asked to wear blinded continuous glucose monitoring device for 14 days.

SUMMARY:
The aim of this study is to determine the ability of postpartum continuous glucose monitoring (CGM) for subjects with gestational diabetes (GDM) to predict dysglycemia on 4-12 week postpartum oral glucose tolerance test (OGTT).

DETAILED DESCRIPTION:
Gestational diabetes (GDM) is glucose intolerance that develops during pregnancy. In the US, GDM affected 8.3% of pregnancies in 2021. Persistent glucose intolerance is present in up to 20% of women at post-partum follow up and subsequent risk for type 2 diabetes is significantly increased. All patients with GDM should undergo post-partum oral glucose tolerance test (OGTT) at 4-12 weeks to identify persistence glucose intolerance or overt diabetes. Detecting postpartum dysglycemia in people with GDM is a critical step for reducing long-term risk of type 2 diabetes and its associated complications. However, <50% of people complete the postpartum OGTT due to barriers in transportation, finances, and childcare. Recent studies have examined the use of postpartum continuous glucose monitoring (CGM) and proposed CGM metrics to predict dysglycemia on postpartum OGTT in people with GDM. These findings should be validated in other cohorts to confirm broad applicability.

This pilot study aims to enroll subjects with GDM at the University of Chicago to wear a blinded CGM for 14 days postpartum (study intervention) and then complete a OGTT at 4-12 weeks postpartum (standard of care).

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18
2. Completed pregnancy with delivery of a live born infant(s). Pregnancies with multiple gestations will be included
3. No prior history of type 1 or type 2 diabetes

   * Patients with a history of gestational diabetes (GDM) in a prior pregnancy will be eligible for inclusion.
4. GDM diagnosis by standard screening at 24-28 weeks

   * 2 hour 75g oral glucose tolerance test (OGTT); one abnormal value required for diagnosis

     * Fasting glucose 92
     * 1 hour 180
     * 2 hour 153
   * 3 hour 100g OGTT - two abnormal values required for diagnosis

     * Fasting glucose - 95
     * 1 hour 180
     * 2 hour 155
     * 3 hour 140

There are no exclusion criteria for this study. Eligibility will be based on inclusion criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Determine the ability of continuous glucose monitoring to predict dysglycemia | baseline to Day 70
  Assess the validity of the continuous glucose monitoring metrics (percentage) proposed by Cabrera et al. (percent time >180 of >4%)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Dickens, MD, Principal Investigator — University of Chicago

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] QuickStats: Percentage of Mothers with Gestational Diabetes,* by Maternal Age - National Vital Statistics System, United States, 2016 and 2021. MMWR Morb Mortal Wkly Rep. 2023 Jan 6;72(1):16. doi: 10.15585/mmwr.mm7201a4. No abstract available. PMID 36602935
- [Background] Kjos SL, Buchanan TA, Greenspoon JS, Montoro M, Bernstein GS, Mestman JH. Gestational diabetes mellitus: the prevalence of glucose intolerance and diabetes mellitus in the first two months post partum. Am J Obstet Gynecol. 1990 Jul;163(1 Pt 1):93-8. doi: 10.1016/s0002-9378(11)90676-0. PMID 2375376
- [Background] Catalano PM, Vargo KM, Bernstein IM, Amini SB. Incidence and risk factors associated with abnormal postpartum glucose tolerance in women with gestational diabetes. Am J Obstet Gynecol. 1991 Oct;165(4 Pt 1):914-9. doi: 10.1016/0002-9378(91)90438-w. PMID 1951553
- [Background] American Diabetes Association Professional Practice Committee. 15. Management of Diabetes in Pregnancy: Standards of Care in Diabetes-2025. Diabetes Care. 2025 Jan 1;48(1 Suppl 1):S306-S320. doi: 10.2337/dc25-S015. PMID 39651985
- [Background] Werner EF, Has P, Kanno L, Sullivan A, Clark MA. Barriers to Postpartum Glucose Testing in Women with Gestational Diabetes Mellitus. Am J Perinatol. 2019 Jan;36(2):212-218. doi: 10.1055/s-0038-1667290. Epub 2018 Jul 30. PMID 30060291
- [Background] Cabrera C et al. Postpartum Dysglycemia Screening with Continuous Glucose Monitoring. Diabetes 2024;73(Supplement_1):1973-LB